CLINICAL TRIAL: NCT06245551
Title: A Phase III, Multicentre, Randomized, Double-blind, Single-Dose, 2-Arm, 2-Period, Crossover Study to Investigate the Efficacy of PT027 Compared With Placebo on Exercise-Induced Bronchoconstriction in Adult Patients With Asthma (BREATH)
Brief Title: A Study to Investigate the Effects of PT027 (Budesonide/Albuterol Sulfate) Metered-dose Inhaler Compared With Placebo on Exercise-Induced Bronchoconstriction in Adult Patients With Asthma
Acronym: BREATH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZ-RU-00004
Record Dates: First submitted 2023-12-13; First posted 2024-02-07 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Asthma, Exercise-Induced
Keywords: Asthma; Exercise-Induced Allergies; Bronchial Spasm; Albuterol; Budesonide; Bronchodilator Agents; Anti-Inflammatory Agents
MeSH Terms: conditions — Asthma, Exercise-Induced; Asthma; Exercise-Induced Allergies; Bronchial Spasm | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- A/B - Treatment with PT027 (BUDESONIDE/ALBUTEROL) 160/180 μg followed by treatment with Placebo (Experimental): Subjects randomized to receive a single dose of PT027 160/180 μg in treatment Period 1, and a single dose of Placebo in treatment Period 2.
  Interventions: Drug: Budesonide/albuterol metered-dose inhaler 160/180 μg; Drug: Placebo metered-dose inhaler
- B/A - Treatment with Placebo followed by treatment with PT027 (BUDESONIDE/ALBUTEROL) 160/180 μg (Experimental): Subjects randomized to receive a single dose of Placebo in treatment Period 1, and a single dose of PT027 160/180 in treatment Period 2.
  Interventions: Drug: Budesonide/albuterol metered-dose inhaler 160/180 μg; Drug: Placebo metered-dose inhaler

INTERVENTIONS:
Drug: Budesonide/albuterol metered-dose inhaler 160/180 μg — Budesonide/albuterol combination aerosol for inhalation, single dose (given as 2 actuations of 80/90 μg)
  Other Names: PT027 (BDA MDI) 160/180 μg
Drug: Placebo metered-dose inhaler — Placebo aerosol for inhalation, single dose (given as 2 actuations)
  Other Names: Placebo MDI

SUMMARY:
The purpose of this Phase III, multicentre, randomized, double-blind, single-dose, 2-period, crossover study is to assess the efficacy and safety of PT027 (budesonide/albuterol sulfate) metered-dose inhaler compared with placebo on exercise-induced bronchoconstriction in adult patients with asthma. Subjects will receive each study treatment on separate visits and undergo a treadmill exercise challenge test so that the effect of study treatment on exercise-induced bronchoconstriction can be evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged 18 to 70 years at the time of informed consent.
2. Documented history of asthma for at least 6 months prior to Visit 1
3. Receiving 1 of the following asthma therapies with stable dosing for at least the 4 weeks before Visit 1 (no other asthma therapies are permitted during the study):

   * Short-acting β 2-adrenoreceptor agonist (SABA) used as needed;
   * Low- to medium-dose maintenance therapy with inhaled corticosteroid (ICS) and SABA used as needed.
4. Demonstrate acceptable MDI administration technique (use of a spacer device during the treatment phase is not permitted)

Exclusion Criteria:

1. Chronic obstructive pulmonary disease or other significant lung disease (eg, chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, bronchopulmonary dysplasia), including regular or occasional use of oxygen.
2. Systemic corticosteroids (SCS) use (any dose and any indication) within 3 months before Visit 1.
3. History of life-threatening asthma, defined by past intubations for asthma, or intensive care unit admission for asthma within the prior 24 months.
4. Receiving regular maintenance treatment with prohibited anti-inflammatory or long-acting bronchodilator asthma medication (inhaled, nebulized, oral, or systemic) within 1 month prior to Visit 1.
5. Unable to tolerate the lung function testing performed after exercise challenge test without use of rescue medication.
6. Current smokers, former smokers with >10 pack-years history, or former smokers who stopped smoking <6 months before Visit 1 (including all forms of tobacco, e-cigarettes [vaping], and marijuana).
7. Completed treatment for lower respiratory infection within 6 weeks prior to Visit 1, regardless if resulting in accompanying asthma symptoms aggravation or not.
8. Upper respiratory infection involving antibiotic treatment not resolved within 7 days prior to Visit 1.
9. Received any marketed (eg, omalizumab, mepolizumab, reslizumab, benralizumab, dupilumab) or investigational biologic within 3 months before Visit 1, or any other prohibited medication.
10. Historical or current evidence of a clinically significant disease.
11. History of psychiatric disease or intellectual deficiency.
12. Having a scheduled or planned hospitalization during the study.
13. Inability (and/or unwillingness) to abstain from protocol-defined prohibited medications during the study.
14. Use of any herbal products by inhalation or nebulizer within 2 weeks of Visit 1 and/or the unwillingness to stop during the study duration.
15. Significant abuse of alcohol or drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - Research Site, Moscow
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Ulyanovsk

REFERENCES:
- See also: AZ-RU-00004_CSP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=AZ-RU-00004&attachmentIdentifier=8eabc9e6-e53d-4c17-aaae-9b10b2e08ce2&fileName=AZ-RU-00004_CSP_Redacted.pdf&versionIdentifier=
- See also: AZ-RU-00004_Statistical Analysis Plan_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=AZ-RU-00004&attachmentIdentifier=ae80b3f5-d4df-40a3-9541-335da5e4ba22&fileName=AZ-RU-00004_Statistical_Analysis_Plan_Redacted.pdf&versionIdentifier=
- See also: AZ-RU-00004_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=AZ-RU-00004&attachmentIdentifier=60ac9ac9-d79d-4285-a0da-81c01107d24c&fileName=AZ-RU-00004_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Budesonide/Albuterol Metered-dose Inhaler (BDA MDI) 160/180 - Placebo: Participants administered BDA MDI 160/180 during 1st period and placebo in 2nd period
- Placebo - Budesonide/Albuterol Metered-dose Inhaler (BDA MDI) 160/180: Participants administered placebo during 1st period and BDA MDI 160/180 in 2nd period
Period: Overall Study
Arm/Group | Budesonide/Albuterol Metered-dose Inhaler (BDA MDI) 160/180 - Placebo | Placebo - Budesonide/Albuterol Metered-dose Inhaler (BDA MDI) 160/180
Started | 31 | 33
Completed | 31 | 33
Not Completed | 0 | 0
Period: 1st Period
Arm/Group | Budesonide/Albuterol Metered-dose Inhaler (BDA MDI) 160/180 - Placebo | Placebo - Budesonide/Albuterol Metered-dose Inhaler (BDA MDI) 160/180
Started | 31 | 33
Completed | 31 | 33
Not Completed | 0 | 0
Period: 2nd Period
Arm/Group | Budesonide/Albuterol Metered-dose Inhaler (BDA MDI) 160/180 - Placebo | Placebo - Budesonide/Albuterol Metered-dose Inhaler (BDA MDI) 160/180
Started | 31 | 33
Completed | 31 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide/Albuterol Metered-dose Inhaler (BDA MDI) 160/180 - Placebo | Placebo - Budesonide/Albuterol Metered-dose Inhaler (BDA MDI) 160/180 | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (14.5) | 43.2 (13.9) | 41.1 (14.2)
Age, Customized [Number; unit: Participants]
  < 65 years | 30 | 32 | 62
  >= 65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 12 | 16 | 28
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 31 | 33 | 64
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 32 | 63
  Not Reported | 0 | 1 | 1
Pre-dose pre-exercise challenge test (ECT) forced expiratory volume in 1 second (FEV1) [Mean (Standard Deviation); unit: liters] | 2.925 (0.826) | 3.042 (0.877) | 2.985 (0.848)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percentage Fall From Post-dose, Pre-exercise Baseline in Forced Expiratory Volume in 1 Second (FEV₁) Observed up to 60 Minutes Post-exercise Challenge
Description: Lung function was measured by spirometry. Spirometry assessments were completed 5 minutes before dosing, 30 minutes after dosing (baseline; 5 minutes before the exercise challenge), and then 5, 10, 15, 30, and 60 minutes after the exercise challenge. A reduction in FEV₁ was expected due to the effects of asthma and exercise on breathing and lung function. The percentage fall in FEV₁ was calculated based on the baseline value and maximum percentage fall value during the 60-minute assessment period.
Time Frame: Up to 60 minutes post-exercise challenge
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent fall
Groups:
- BDA MDI 160/180: Participants administered BDA MDI 160/180 during 1st or 2nd period
- Placebo: Participants administered placebo during 1st or 2nd period
Arm/Group | BDA MDI 160/180 | Placebo
Number analyzed (Participants) | 64 | 64
Percent fall
  All subjects | 6.95 [5.36 to 8.54] | 24.46 [22.87 to 26.05]
  Non-ICS: number analyzed (Participants) | 23 | 23
  Non-ICS | 6.28 [3.63 to 8.93] | 26.62 [23.97 to 29.28]
  ICS: number analyzed (Participants) | 41 | 41
  ICS | 7.29 [5.32 to 9.25] | 23.28 [21.32 to 25.25]
Statistical Analysis 1: Comparison: BDA MDI 160/180 vs Placebo; Test type: Other — The analysis is applied to the All-subjects data; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -17.52, 95% CI 2-sided [-19.78 to -15.25]

2. Secondary Outcome: Percentage of Subjects With a Maximum Percentage Fall in FEV₁ Post-exercise Challenge of <10% and <20%
Description: The percentage fall in FEV₁ was calculated based on the baseline value and maximum percentage fall value during the 60-minute assessment period, and the percentage of subjects with a maximum percentage fall <10% and <20% was determined
Time Frame: Up to 60 minutes post exercise challenge
Measure: Count of Participants; unit: Participants
Arm/Group | BDA MDI 160/180 | Placebo
Number analyzed (Participants) | 64 | 64
Participants
  Maximum percentage fall <10% | 48 | 2
  Maximum percentage fall <20% | 62 | 14

3. Secondary Outcome: Percentage Fall From Post-dose, Pre-exercise Baseline in FEV1 at Each Time Point Within 60 Minutes Post-exercise Challenge
Description: The percentage fall in FEV₁ at each time point was calculated based on the baseline value and percentage fall value during the 60-minute assessment period at each time point.
Time Frame: Up to 60 minutes post exercise challenge
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | BDA MDI 160/180 | Placebo
Number analyzed (Participants) | 64 | 64
Percent
  5 min Post-ECT | 1.68 [-0.11 to 3.47] | 9.79 [8.00 to 11.58]
  10 min Post-ECT | 3.16 [1.30 to 5.02] | 17.98 [16.12 to 19.84]
  15 min Post-ECT | 4.20 [2.38 to 6.03] | 19.14 [17.31 to 20.97]
  30 min Post-ECT | 2.64 [0.65 to 4.63] | 11.85 [9.87 to 13.84]
  60 min Post-ECT | 0.56 [-0.83 to 1.94] | 3.10 [1.72 to 4.48]

4. Secondary Outcome: Post-Exercise FEV1 Area Under the Curve From 0 to 30 Minutes (AUC0-30min)
Description: FEV1 AUC0-30min will be derived for the changes from the post-dose, pre-exercise baseline using the trapezoidal rule and will be normalized by dividing by the actual time (in minutes) from dosing to the last included measurement, scheduled at 30 minutes post-exercise challenge.
Time Frame: Up to 30 minutes post exercise challenge
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | BDA MDI 160/180 | Placebo
Number analyzed (Participants) | 64 | 64
liter | -0.10 (0.16) | -0.44 (0.23)

5. Secondary Outcome: Time To Recovery
Description: Time to recovery will be derived as the time (minutes) post-exercise challenge in which the FEV1 result returns to within 10% of the value recorded at the post-dose, pre-exercise baseline.
Time Frame: Up to 60 minutes post exercise challenge
Measure: Count of Participants; unit: Participants
Arm/Group | BDA MDI 160/180 | Placebo
Number analyzed (Participants) | 64 | 64
Participants | 56 | 6

6. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs)
Description: The safety profile will be evaluated using vital signs, physical examination, electrocardiograms (ECGs) and AE data.
Time Frame: Through study completion, an average of 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BDA MDI 160/180 | Placebo
Number analyzed (Participants) | 64 | 64
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse events presented in the tables below were collected during up to 19 days from the time of first study treatment to follow-up telephone call. Actual time for each participant depends on duration of their participation in the study.
Arm/Group | BDA MDI 160/180 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 1/64 | 2/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BDA MDI 160/180 (N=64) | Placebo (N=64)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Bronchial irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT06245551/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT06245551/SAP_001.pdf